CLINICAL TRIAL: NCT07263503
Title: Clip and Coil: A Novel Safe Strategy in Managing Fundal Gastric Varices With a Large Spontaneous Portosystemic Shunt
Brief Title: Clip and Coil in Fundal Gastric Varices With a Large Shunt
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-1588
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Fundal Gastric Varices; Endoscopic Ultrasound (EUS)-Guided Coil Deployment; Titanium Clips; Ectopic Embolization; Gastric Variceal Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fundal gastric varices associated with a large spontaneous portosystemic shunt (>1cm): Clips were placed before EUS-guided coil deployment

SUMMARY:
Endoscopic ultrasound (EUS)-guided coil deployment is a promising technique for the endoscopic management of gastric varices. However, coil migration may occur in patients with large drainage collaterals. This study aimed to evaluate the safety and efficacy of using clips in combination with coils for treating gastric varices. In this retrospective study, clips were placed before EUS-guided coil deployment in each patient with gastric varices and a large spontaneous portosystemic shunt. The pressure of gastric varices was directly measured by puncturing the varix with a needle connected to a pressure transducer, before and after clip placement. The occurrence of ectopic embolization or coil migration was recorded.

ELIGIBILITY:
Inclusion Criteria:

1. presence of a spontaneous portosystemic shunt, including gastrorenal or splenorenal collateral shunts;
2. use of both clips and coils during endoscopic intervention.

Exclusion Criteria:

The spontaneous portosystemic shunt was narrow (diameter < 1.0 cm).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with fundal gastric varices, admitted for endoscopic intervention
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The occurrence of ectopic embolization | Within the day of the endoscopic intervention (after the operation)

SECONDARY OUTCOMES:
The occurrence of coil migration | Within the day of the endoscopic intervention (after the operation)

OTHER OUTCOMES:
Gastric variceal pressure gradient | During the endoscopic intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No